CLINICAL TRIAL: NCT01763580
Title: Open-Label, Randomized, Comparative, Multi-Center Clinical Trial on the Therapeutic Effect of Tacrolimus (Prograf Cap.®) in Combination With Low-Dose Corticosteroid Compared With High-Dose Corticosteroid Alone in Patients With Minimal-Change Nephrotic Syndrome (MCNS)
Brief Title: A Study to Evaluate the Effect of Tacrolimus and Corticosteroid Combination Therapy in Patients With Minimal Change Nephrotic Syndrome
Acronym: T-OPTIMUM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRGNS-11-02-KOR
Record Dates: First submitted 2012-12-06; First posted 2013-01-09 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: MCNS; Minimal Change Nephrotic Syndrome (MCNS)
Keywords: Glomerulonephritis; Tacrolimus; Nephrotic syndrome
MeSH Terms: conditions — Nephrosis, Lipoid; Glomerulonephritis; Nephrotic Syndrome | interventions — Tacrolimus; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tacrolimus with low-dose corticosteroid (Experimental): Oral
  Interventions: Drug: Tacrolimus; Drug: Prednisolone
- High-dose corticosteroid alone (Active Comparator): Oral
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Tacrolimus — Oral
  Other Names: FK506; Prograf Capsule
  Arms: Tacrolimus with low-dose corticosteroid
Drug: Prednisolone — Oral

SUMMARY:
To compare the therapeutic effect of tacrolimus in combination with low-dose corticosteroid with high-dose corticosteroid alone in patients with minimal-change nephrotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been diagnosed with initial or relapsed primary minimal-change nephrotic syndrome
* patients whose urine protein-creatinine ratio (UPCR) is more than 3.0

Exclusion Criteria:

* patients whose eGFR is less than 30 ml/min/1.73 m2
* patients who were treated with immunosuppressants, such as tacrolimus, cyclosporine, cyclophosphamide (Cytoxan), mizoribine (Bredinin), levamisole, azathioprine, mycophenolate mofetil, or rituximab, within two weeks before the study
* patients to whom more than 10 mg prednisolone or an equivalent dose of steroid was administered daily within two weeks before the study
* patients who are pregnant, breastfeeding, or planning to be pregnant or to breastfeed within six months after the study completion, or who cannot or do not want to use any contraceptive method
* patients who are hypersensitive to the investigational drug or to macrolide, such as azithromycin, clarithromycin, or roxithromycin
* patients who were treated with a live vaccine within four weeks before the study
* patients whose liver panel laboratory test result is three times the normal range, or acute hepatitis patients whose serum bilirubin has been clinically significantly higher than 3.6 mg/dL for more than 1 month
* patients who have a significant general disease that makes it inappropriate for them to participate in this study as adjudged by the investigator (e.g., cardiovascular-acute myocardial infarction, heart failure [classified as more than New York Heart Association {NYHA} class III], hepatic/gastrointestinal/neurologic disease, blood disorder, cancer, infection, renal disorder other than minimal-change nephrotic syndrome, rheumatic arthritis with pneumonia interstitials)
* patients who have genetic problems such as galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption
* patients to whom another investigational drug was administered within 30 days from the enrollment in the study
* patients who participated in the past phases of this study

Ages: 16 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2012-07-16 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-08-21 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects who show a decreased UPCR (Urine Protein Creatinine Rate) of less than 0.2 | up to 8 weeks after treatment

SECONDARY OUTCOMES:
The period until the UPCR is decreased below 0.2 | up to 8 weeks after treatment
The percentage of subjects who show relapse after the remission | up to 24 weeks
The period until the relapse happens from the complete remission | up to 24 weeks
Safety assessed by the incidence of adverse events, labo-tests, vital signs, ECGs and chest X-rays | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Azukaitis K, Palmer SC, Strippoli GF, Hodson EM. Interventions for minimal change disease in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2022 Mar 1;3(3):CD001537. doi: 10.1002/14651858.CD001537.pub5. PMID 35230699
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=257